CLINICAL TRIAL: NCT02394730
Title: A Double Blind Randomised Comparison of Vorapaxar Versus Placebo for the Treatment of HIV Associated Inflammation and Coagulopathy in Patients With Well Controlled HIV Replication
Brief Title: Attenuation of D-dimer Using Vorapaxar to Target Inflammatory and Coagulation Endpoints
Acronym: ADVICE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Minnesota (Other); University of Melbourne (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-01-ADV; AI000585-26-288416 (Other: NIAID)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: HIV
Keywords: HIV, d-dimer, hs-CRP, activated T-lymphocytes
MeSH Terms: interventions — vorapaxar; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vorapaxar (Experimental): 2.5mg of vorapaxar po qd
  Interventions: Drug: vorapaxar
- Placebo (Placebo Comparator): sugar pill po qd
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vorapaxar — 2.5mg of vorapaxar taken orally once daily for 12 weeks
  Other Names: Zontivity
  Arms: vorapaxar
Drug: Placebo — Sugar pill taken orally once daily for 12 weeks
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
ADVICE is a randomised, international, double-blind, placebo-controlled trial. The purpose of the ADVICE study is to compare the safety and efficacy of vorapaxar in reducing d-dimer expression and markers of cellular immune activation over a period of 12 weeks among people with HIV infection who are successfully treated with combination antiretroviral therapy containing an HIV integrase inhibitor. A secondary objective of the study will be to demonstrate that following cessation of vorapaxar in patients with well controlled HIV replication there will be an increase in the levels of d-dimer over a 6 week period. 60 participants from 4 clinical sites in Australia and the USA will be recruited and followed for a minimum of 18 weeks.

DETAILED DESCRIPTION:
Consenting participants will be screened and within 14 days randomly allocated to receive either vorapaxar (2.5mg) or matched placebo once daily for 12 weeks (phase 1). Participants will be seen one week after randomisation and then at weeks 4, 8 and 12 (phase 1). At the week 12 visit, patients will not be dispensed any study treatment. In phase 2 all study treatment will stop for 6 weeks. At week 18 patients will be seen for a final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive by licensed diagnostic test
2. aged ≥40 years
3. plasma HIV RNA <50 copies/mL for at least 24 weeks
4. screening CD4+ cell count > 50 cells/mm3
5. treated for at least 12 weeks with a suppressive regimen of combination antiretroviral therapy that does not include HIV protease inhibitors and/or NNRTIs (except rilpivirine)
6. plasma d-dimer >200ng/mL (>0.2μg/mL or >0.2mg/L) fibrinogen equivalent units or >100ng/mL (>0.1 μg/mL or >0.1mg/L) d-dimer units in the absence of established cause (deep vein thrombosis/embolism)
7. provision of written informed consent

Exclusion Criteria:

1. Absolute neutrophil count (ANC) <1000 cells/μL
2. hemoglobin <10.0 g/dL
3. platelet count <75,000 cells/μL
4. AST and/or ALT >2.5 x ULN
5. estimated glomerular filtration rate <30mL/min/1.73m2 ) using CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation
6. history of myocardial infarction or unstable atherosclerotic disease
7. history of ischemic stroke or transient ischaemic attack (TIA)
8. active peptic/duodenal ulcer or other bleeding disorder within the previous 12 months
9. intent to have surgery within the 6 month period after randomisation
10. current use of aspirin or P2Y12 antiplatelet therapy
11. use of anticoagulants, (eg. heparin or warfarin), fibrinolytic therapy, chronic use (more than 5 consecutive days) of nonsteroidal anti-inflammatory drugs (NSAIDS), strong CYP3A4 inhibitors or inducers. See Manual of Operations for full list of medications to avoid.
12. participants unlikely to be able to remain in follow-up
13. pregnant or nursing mothers
14. in the clinical judgement of the investigator, participation in this trial is deemed inappropriate as this may conflict with the well-being of the participant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Emery, Study Director — University of NSW, Kirby Institute
Locations (7):
- United States (2):
  - Georgetown University Hospital, Georgetown, Maryland
  - Hennepin County Medical Centre, Minneapolis, Minnesota
- Australia (5):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Northside Clinic, Fitzroy North, Victoria
  - Monash Medical Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] ADVICE study group. Vorapaxar for HIV-associated inflammation and coagulopathy (ADVICE): a randomised, double-blind, placebo-controlled trial. Lancet HIV. 2018 Oct;5(10):e553-e559. doi: 10.1016/S2352-3018(18)30214-5. Epub 2018 Sep 23. PMID 30257802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and randomised from 2 sites in USA and 5 sites in Australia.
Pre-assignment Details: 125 were screened and 60 were not randomised (55 ineligible, 4 lost to follow up and 1 withdrew consent prior to randomisation).
Period: Overall Study
Arm/Group | Vorapaxar | Placebo
Started | 34 | 31
Completed | 33 | 30
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant was lost to follow up immediately after randomisation and did not receive a single dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorapaxar | Placebo | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [48 to 58] | 52 [48 to 60] | 52 [48 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 31 | 28 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 23 | 48
  Asian | 1 | 2 | 3
  Black | 7 | 5 | 12
  Hispanic/Latino | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
  Australia | 21 | 21 | 42
Total Cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 4.6 [4.0 to 5.5] | 4.7 [3.9 to 5.4] | 4.7 [4.0 to 5.4]
HDL Cholesterol [Median (Inter-Quartile Range); unit: (mmol/L)] | 1.2 [1.0 to 1.4] | 1.3 [0.9 to 1.6] | 1.2 [1 to 1.5]
Systolic blood pressure [Median (Inter-Quartile Range); unit: (mm Hg)] | 125 [115 to 133] | 127 [120 to 136] | 126.5 [117.5 to 135]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: (mm Hg)] | 77 [70 to 85] | 80 [70 to 86] | 78.5 [70 to 85.5]
Current smoker [Count of Participants; unit: Participants] | 9 | 9 | 18
Framingham 10 yr CHD Risk Score [Median (Inter-Quartile Range); unit: Percentage of risk] — Framingham Heart Score: 10 year Coronary Heart Disease Risk Score was calculated at baseline using methods published by D'Agostino. Factors including age, sex, smoking status, Total Cholesterol, HDL Cholesterol, systolic blood pressure, treatment for blood pressure.
  Percentage of risk | 10.6 [7.3 to 21.1] | 12.1 [8.3 to 19.4] | 11.4 [7.9 to 19.8]
d-dimer [Median (Inter-Quartile Range); unit: ng/mL] | 432.5 [298 to 531.1] | 391.6 [302.3 to 813.7] | 421.9 [299 to 687.6]
High sensitivity C Reactive Protein (hs-CRP) [Median (Inter-Quartile Range); unit: ug/mL] | 1.53 [0.50 to 3.01] | 1.97 [0.61 to 4.81] | 1.58 [0.50 to 3.86]
Interleukin 6 (IL-6) [Median (Inter-Quartile Range); unit: pg/mL] | 0.93 [0.61 to 1.39] | 0.99 [0.69 to 1.54] | 0.94 [0.62 to 1.52]
Estimated duration of HIV infection [Median (Inter-Quartile Range); unit: years] | 12.8 [9.2 to 24.3] | 12.2 [8.6 to 22.4] | 12.5 [8.8 to 23.2]
Plasma HIV RNA [Median (Inter-Quartile Range); unit: copies/mL] | 20 [20 to 48] | 20 [20 to 48] | 20 [20 to 48]
CD4 count [Median (Inter-Quartile Range); unit: cells per uL] | 639 [504 to 768] | 698 [490 to 869] | 643 [497 to 829]
Time on current Anti-Retroviral Treatment regimen [Median (Inter-Quartile Range); unit: years] | 1.3 [0.7 to 3] | 2 [0.7 to 4] | 1.5 [0.7 to 3.9]

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline for D-dimer (ng/mL) to the Average of Weeks 8 and 12
Description: Mean of week 8 and week 12 minus week 0 (on log10 scale) then back transforming the log10 difference to obtain percentage change from baseline.
Time Frame: at week 8 and week 12
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 31
percent | -10.8 [-23.1 to 3.4] | -8.5 [-18.4 to 2.5]

2. Secondary Outcome: Number of Participants in Each Treatment Group With Plasma HIV-1 RNA <50 Copies/mL
Description: Number of participants in each treatment group with plasma HIV-1 RNA <50 copies/mL at week 18
Time Frame: at week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
Participants | 31 | 29

3. Secondary Outcome: Mean Change From Baseline to Week 12 in CD4+ Cell Counts
Description: Mean of week 12 CD4+ cell count minus mean of week 0 CD4+ cell count
Time Frame: at week 12
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 29 | 28
cells/mm3 | -21.3 (143.7) | -29.7 (400.3)

4. Secondary Outcome: Mean Change From Baseline to Week 12 in CD8+ Cell Counts
Description: Mean of week 12 CD8+ cell count minus mean of week 0 CD4+ cell count
Time Frame: at week 12
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 29 | 28
cells/mm3 | 3 (191.6) | 81.1 (244.7)

5. Secondary Outcome: Number of Patients in Each Treatment Group With D-dimer <165ng/mL at Week 12
Description: Number of patients in each treatment group with d-dimer <165ng/mL at week 12
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
Participants | 1 | 2

6. Secondary Outcome: Number of Patients in Each Treatment Group With D-dimer > or Equal to 165ng/mL at Week 18
Description: Number of patients in each treatment group with d-dimer > or equal to 165ng/mL at week 18
Time Frame: week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
Participants | 32 | 29

7. Secondary Outcome: Mean Change From Baseline in log10 D-Dimer
Description: Differences between treatment groups in mean change from week 0 log10 d-dimer to week 18
Time Frame: at week 18
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
percent change | -2.21 [-17.9 to 16.5] | -14.1 [-17.7 to 17.9]

8. Secondary Outcome: Mean Change From Baseline in log10 Hs-CRP at Week 18
Description: Differences between treatment groups in mean change from baseline log10 hs-CRP to week 18. ie Week 18 log10 hs-CRP minus week 0 log10 hs-CRP
Time Frame: at week 18
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
pg/mL | -0.03 (0.39) | -0.10 (0.54)

9. Secondary Outcome: Percent Change From Baseline Hs-CRP (ug/mL) to the Average of Week 8 and Week 12
Description: Mean of week 8 and week 12 minus week 0 (on log10 scale) then back transformed the log10 difference to obtain percentage change from baseline.
Time Frame: week 8 and 12
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
Percent | -0.02 [-41.3 to 70.2] | -15.7 [-40.9 to 20.2]

10. Secondary Outcome: Mean Percent Change From Baseline IL-6 (pg/mL) to the Average of Week 8 and Week 12
Description: as for outcome 9
Time Frame: at week 8 and week 12
Measure: Mean (90% Confidence Interval); unit: percent
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
percent | 12.6 [-15.6 to 50.4] | -11.6 [-29.1 to 10.3]

11. Secondary Outcome: Differences Between Treatment Groups in Mean Change From Baseline log10 IL-6
Description: Differences between treatment groups in mean change from baseline log10 IL-6 at week 18
Time Frame: at week 18
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 30
pg/mL | 0.03 (0.36) | -0.10 (0.25)

12. Secondary Outcome: Total Number of Participants With BARC Type 1, 2, 3, 4, or 5 Bleeding Episodes
Description: Bleeding Academic Research Consortium (BARC) Definitions for Bleeding Events Type 1 -bleeding that is not actionable and does not cause the patient to seek unscheduled performance of studies, hospitalization, or treatment by a healthcare professional; may include episodes leading to self-discontinuation of medical therapy by the patient without consulting a healthcare professional Type 2 - overt, actionable sign of haemorrhage (eg, more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for type 3, 4, or 5 but does meet at least one of the following criteria: (1) requiring nonsurgical, medical intervention by a healthcare professional, (2) leading to hospitalization or increased level of care, or (3) prompting evaluation Type 3- Bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid) Type 4 - Coronary Artery Bypass Graft procedure-related bleeding Type 5 -
Time Frame: at week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 31
Participants | 12 | 10

13. Secondary Outcome: Total Number of Participants With Any SAE Between Baseline and Week 18
Description: Total number of participants with any SAE between baseline and week 18
Time Frame: week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 31
Participants | 3 | 2

14. Secondary Outcome: Total Number of Participants With Any AE Between Baseline to Week 18
Description: Total number of participants with any AE between week 0 to week 18
Time Frame: week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 33 | 31
Participants | 28 | 28

15. Secondary Outcome: Changes From Baseline in Renal Function Measured by the CKD-EPI Estimate of Creatinine Clearance at Week 12
Description: Changes from baseline in renal function measured by the CKD-EPI estimate of creatinine clearance at week 12
Time Frame: at week 12
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 31 | 30
ml/min/1.73m2 | 2.08 (8.38) | 2.05 (7.71)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Vorapaxar | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/33 | 2/31
Other Adverse Events (participants affected / at risk) | 15/33 | 22/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar (N=33) | Placebo (N=31)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
spinal stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Post Procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar (N=33) | Placebo (N=31)
Upper Respiratory Tract Injection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (8)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Epistaxis (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Contusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Pain in extremety (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peripheral Swelling (General disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators need to submit a proposal, abstract, manuscript or other form of communication of trial results to the Protocol Steering Committee for review and approval.

DOCUMENTS (2):
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT02394730/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT02394730/SAP_001.pdf